CLINICAL TRIAL: NCT01390220
Title: A Randomized, Double-blind, Placebo-controlled Study of the Safety and Efficacy of Intranasal Midazolam (USL261) in the Outpatient Treatment of Subjects With Seizure Clusters. ARTEMIS-1: Acute Rescue Therapy in Epilepsy With Midazolam Intranasal Spray-1
Brief Title: Study to Evaluate the Safety and Efficacy of USL261 (Intranasal Midazolam) in Patients With Seizure Clusters
Acronym: ARTEMIS1
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma S.P.R.L. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P261-401; 2011-001318-32 (EudraCT Number)
Record Dates: First submitted 2011-07-06; First posted 2011-07-08 (Estimated); Results first posted 2019-05-31 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Epilepsy
Keywords: Epilepsy; seizure clusters; acute repetitive seizures; rescue treatment; ARTEMIS
MeSH Terms: conditions — Epilepsy; Severe combined immunodeficiency with sensitivity to ionizing radiation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- USL261 (Experimental): intranasal midazolam 5mg
  Interventions: Drug: USL261
- Placebo (Experimental): Intranasal placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: USL261
  Other Names: Midazolam nasal spray (MDZ NS)
  Arms: USL261
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the safety and effectiveness of USL261 for the outpatient treatment of seizure clusters.

DETAILED DESCRIPTION:
Qualifying participants underwent an in-clinic administration (Test Dose Phase [TDP]) of two doses of USL261 (intranasal midazolam 5 mg), separated by 10 minutes, in the absence of seizures. Eligible participants were then randomized to USL261 versus Placebo in an outpatient Comparative Phase (CP). When the participant had a qualifying seizure cluster episode, as described in an individualized patient management plan, the participant's caregiver administered the double-blind dose. An open-label USL261 dose could be administered after 10 minutes and up to 6 hours after the double-blind dose, if the participant had persistent or recurrent seizures. Initial participants could not proceed to CP until an independent data safety monitoring board (DSMB) reviewed safety data from at least the first 25 participants in TDP; the DSMB performed additional safety reviews at pre-set intervals based on enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Has a competent, adult caregiver who can recognize and observe the subject's seizure cluster episodes
* Has an established diagnosis of partial or generalized epilepsy that includes the following:

  * A documented history of seizure clusters lasting a minimum of 10 minutes
  * Seizure cluster pattern is observable, stereotyped, and recognizably different from the subject's other non-cluster seizure activity (if any)
  * A second seizure in the seizure cluster typically occurring within 6 hours from the time of cluster recognition
  * A seizure cluster pattern composed of multiple (≥ 2) partial or generalized seizures
  * A seizure cluster pattern established > 3 months before Visit 1
  * A frequency of ≥ 3 seizure clusters during the year before Visit 1
  * At least 1 seizure cluster occurring ≤ 4 months before Visit 1
  * Seizure cluster pattern is confirmed by a central reviewer
* Currently on a stable regimen of anti-epileptic drugs (AEDs) with no changes in type of AEDs since Visit 1 and for ≥ 7 days before Visit 2, with or without intermittent use of benzodiazepines at a constant dose
* Weight is 40 kg to 125 kg, inclusive

Exclusion Criteria:

* Has a neurological disorder that is likely to progress in the next year
* Has severe chronic cardio-respiratory disease
* Has had psychogenic, non-epileptic seizure(s) within the 5 years before Visit 1
* Has a history of their stereotypical seizure cluster progressing to status epilepticus within the 2 years before Visit 1
* Has a history of acute narrow-angle glaucoma.
* Has had active suicidal plan/intent or active suicidal thoughts in the 6 months before Visit 1 or a suicide attempt in the past 5 years
* Currently using a vagal nerve stimulator (VNS) unless the device has been implanted for at least 6 months and the setting stable for 4 weeks before Visit 1

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (90):
- United States (46):
  - United States, Arizona, Phoenix, Arizona
  - United States, Arizona, Tucson, Arizona
  - United States, Arkansas, Little Rock, Arkansas
  - United States, California, Fresno, California
  - United States, California, Irvine, California
  - United States, California, Loma Linda, California
  - United States, California, Sacramento, California
  - United States, California, Ventura, California
  - United States, Colorado, Aurora, Colorado
  - United States, Connecticut, New Haven, Connecticut
  - United States, Florida, Gainesville, Florida
  - United States, Florida, Gulf Breeze, Florida
  - United States, Florida, Port Charlotte, Florida
  - United States, Florida, Tampa, Florida
  - United States, Florida, Wellington, Florida
  - United States, Idaho, Boise, Idaho
  - United States, Illinois, Chicago, Illinois
  - United States, Kansas, Manhattan, Kansas
  - United States, Kentucky, Lexington, Kentucky
  - United States, Maryland, Baltimore, Maryland
  - United States, Michigan, Detroit, Michigan
  - United States, Minnesota, Saint Paul, Minnesota
  - United States, Missouri, Chesterfield, Missouri
  - United States, Missouri, St Louis, Missouri
  - United States, Nevada, Reno, Nevada
  - United States, New Hampshire, Lebanon, New Hampshire
  - United States, New Jersey, Flemington, New Jersey
  - United States, New Jersey, Hackensack, New Jersey
  - United States, New York, New York, New York
  - United States, New York, Stony Brook, New York
  - United States, New York, The Bronx, New York
  - United States, North Carolina, Durham, North Carolina
  - United States, North Carolina, Winston-Salem, North Carolina
  - United States, Ohio, Columbus, Ohio
  - United States, Oklahoma, Oklahoma City, Oklahoma
  - United States, Oregon, Portland, Oregon
  - United States, Pennsylvania, Philadelphia, Pennsylvania
  - United States, Tennessee, Memphis, Tennessee
  - United States, Tennessee, Nashville, Tennessee
  - United States, Texas, Dallas, Texas
  - United States, Texas, Fort Worth, Texas
  - United States, Texas, Greenville, Texas
  - United States, Texas, San Antonio, Texas
  - United States, Texas, Temple, Texas
  - United States, Virginia, Norfolk, Virginia
  - United States, Wisconsin, Madison, Wisconsin
- Australia (5):
  - Australia, New South Wales, Chatswood, New South Wales
  - Australia, New South Wales, Randwick, New South Wales
  - Australia, Queensland, Herston, Queensland
  - Australia, Vctoria, Heidelberg West, Victoria
  - Australia, Victoria, Parkville, Victoria
- Canada (2):
  - Canada, Ontario, Toronto, Ontario
  - Canada, Quebec, Montreal, Quebec
- Germany (5):
  - Germany, Baden-Wurttemberg, Freiburg im Breisgau, Baden-Wurttemberg
  - Germany, Bayern, Munich, Bavaria
  - Germany, Hessen, Marburg, Hesse
  - Germany, Nordrhein-Westfalen, Bonn, North Rhine-Westphalia
  - Germany, Westfalen-Lippe, Bielefeld, Wetsfalen-Lippe
- Hungary (2):
  - Hungary, Budapest
  - Hungary, Kazincbarcika
- Israel (6):
  - Israel, Haifa
  - Israel, Holon
  - Israel, Jerusalem
  - Israel, Petah Tikva
  - Israel, Ramat Gan
  - Israel, Tel Aviv
- Italy (6):
  - Italy, Florence
  - Italy, Genova
  - Italy, Milan
  - Italy, Napoli
  - Italy, Pavia
  - Italy, San Fermo della Battaglia
- New Zealand (2):
  - New Zealand, Auklund, Grafton, Auklund
  - New Zealand, Canterbury, Christchurch, Canterbury
- Poland (4):
  - Poland, Gdansk
  - Poland, Katowice
  - Poland, Krakow
  - Poland, Olsztyn
- Spain (6):
  - Spain, Andalucia, Seville, Andalusia
  - Spain, Catalonia, Barcelona, Catalonia
  - Spain, Catalonia, Girona, Catalonia
  - Spain, Madrid, Fuencarral-El Pardo, Madrid
  - Spain, Madrid, Moncloa-Aravaca, Madrid
  - Spain, Madrid, Pozuelo de Alarcón, Madrid
- Ukraine (6):
  - Ukraine, Ivano-Frankivsk, Ivano-Frankivsk
  - Ukraine, Kharkiv
  - Ukraine, Odesa
  - Ukraine, Poltava
  - Ukraine, Ternopil
  - Ukraine, Vinnytsia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Meng TC, Szaflarski JP, Chen L, Brunnert M, Campos R, Van Ess P, Pullman WE, Fakhoury T. Psychosocial outcomes of repeated treatment of seizure clusters with midazolam nasal spray: Results of a phase 3, open-label extension trial. Epilepsy Behav. 2023 Jan;138:108989. doi: 10.1016/j.yebeh.2022.108989. Epub 2022 Nov 18. PMID 36410152
- [Derived] Detyniecki K, Van Ess PJ, Sequeira DJ, Wheless JW, Meng TC, Pullman WE. Safety and efficacy of midazolam nasal spray in the outpatient treatment of patients with seizure clusters-a randomized, double-blind, placebo-controlled trial. Epilepsia. 2019 Sep;60(9):1797-1808. doi: 10.1111/epi.15159. Epub 2019 May 29. PMID 31140596

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants underwent in-clinic administration of open-label USL261 5 mg followed by USL261 5 mg 10 minutes in absence of a seizure (Test Dose Phase [TDP]). Participants were then randomized to double-blind USL261 5 mg or Placebo to be administered by caregiver to treat a seizure cluster in Comparative Phase (CP) in the outpatient setting.
Groups:
- USL261 TDP: Participants who received at least 1 open-label USL261 5 mg dose in Test Dose Phase (TDP)
- USL261 CP: Participants completing TDP who received USL261 5 mg as randomized dose to treat a seizure cluster episode in the Comparative Phase (CP)
- Placebo CP: Participants completing TDP who received placebo as randomized dose to treat a seizure cluster episode in the Comparative Phase (CP)
Period: Test Dose Phase
Arm/Group | USL261 TDP | USL261 CP | Placebo CP
Started | 292 | 0 (This arm not applicable in TDP.) | 0 (This arm not applicable in TDP.)
Completed | 201 | 0 | 0
Not Completed | 91 | 0 | 0
Not completed — Adverse Event | 17 | 0 | 0
Not completed — Withdrawal by Subject | 8 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Protocol Violation | 8 | 0 | 0
Not completed — No treated seizure cluster episode | 37 | 0 | 0
Not completed — Study/Site closure | 6 | 0 | 0
Not completed — Caregiver no longer available | 5 | 0 | 0
Not completed — Noncompliance | 2 | 0 | 0
Not completed — Logistical | 6 | 0 | 0
Period: Comparative Phase
Arm/Group | USL261 TDP | USL261 CP | Placebo CP
Started (Patients completing TDP, were randomized, and received double-blind dose in CP) | 0 (This arm not applicable in CP) | 134 | 67
Completed | 0 (This arm not applicable in CP) | 133 | 67
Not Completed | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: USL261 Test Dose: All patients receiving at least 1 dose of USL261 5 mg in TDP.
Groups:
- USL261 Test Dose: Participants who received at least 1 open-label USL261 5 mg dose in Test Dose Phase (TDP)
Arm/Group | USL261 Test Dose
Number analyzed (Participants) | 292
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 18
  Between 18 and 65 years | 272
  >=65 years | 2
Age, Continuous [Median (Full Range); unit: years] | 31.5 [12 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 146
  Male | 146
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22
  Not Hispanic or Latino | 270
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Self reported. Unknown or not reported includes Other, eg. "Slavic".
  Participants
    American Indian or Alaska Native | 2
    Asian | 2
    Native Hawaiian or Other Pacific Islander | 1
    Black or African American | 7
    White | 275
    More than one race | 0
    Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  New Zealand | 1
  Canada | 4
  Hungary | 18
  United States | 118
  Ukraine | 70
  Poland | 14
  Italy | 5
  Israel | 18
  Australia | 19
  Germany | 13
  Spain | 12
Body mass index [Median (Full Range); unit: kg/m^2] — Population: Height not measurable in some patients
  kg/m^2
    number analyzed (Participants) | 287
    (all) | 24.69 [15.8 to 48.5]
Seizure cluster episodes in year before Visit 1 of study [Median (Full Range); unit: seizure cluster episodes] | 15 [3 to 999]
Years had seizure cluster episodes prior to study [Median (Full Range); unit: years] — Population: Unknown or data entered as indefinite (eg >3) for some participants
  years
    number analyzed (Participants) | 283
    (all) | 6.0 [0.3 to 62.0]
Typical number of seizures in seizure cluster episode [Median (Full Range); unit: seizures] — Population: Not reported for 1 subject
  seizures
    number analyzed (Participants) | 291
    (all) | 6.0 [2.0 to 200.0]
Typical duration of seizure cluster episode [Median (Full Range); unit: minutes] — Population: Non-numerical duration (eg "several" hours reported for some participants
  minutes
    number analyzed (Participants) | 278
    (all) | 67.5 [2.5 to 4320.0]

OUTCOME MEASURES:

1. Primary Outcome: Participants Who Met the Criteria for Treatment Success After Administration of the Double-blind Dose in the Comparative Phase (CP)
Description: Treatment Success is defined as achieving both of the following: 1) termination of seizure(s) within 10 minutes after double-blind study drug administration, and 2) no recurrence of seizure(s) beginning 10 minutes after study drug administration to 6 hours after study drug administration. Participants who received the open-label second dose within 6 hours of administration of the double-blind dose were analyzed as having had a seizure.
Time Frame: 6 hours
Population: Randomized participants who received the double-blind dose in the CP.
Measure: Count of Participants; unit: Participants
Groups:
- USL261 CP: 5 mg intranasal midazolam
  USL261
- Placebo CP: Intranasal placebo
  Placebo
Arm/Group | USL261 CP | Placebo CP
Number analyzed (Participants) | 134 | 67
Participants | 72 | 23
Statistical Analysis 1: Comparison: USL261 CP vs Placebo CP; Test type: Superiority; p = 0.0109, Fisher Exact; 2-sided

2. Secondary Outcome: Participants With Seizure(s) >10 Minutes to 4 Hours After Administration of the Double-blind Dose
Description: Participants with recurrence of seizure(s) >10 minutes and up to 4 hours after administration of the double-blind dose in the CP. Participants who received the open-label second dose within 4 hours of administration of the double-blind dose were analyzed as having had a seizure.
Time Frame: 4 hours
Population: Randomized participants who received the double-blind dose in the CP.
Measure: Count of Participants; unit: Participants
Arm/Group | USL261 CP | Placebo CP
Number analyzed (Participants) | 134 | 67
Participants | 51 | 40
Statistical Analysis 1: Comparison: USL261 CP vs Placebo CP; Test type: Superiority; p = 0.0043, Fisher Exact; 2-sided

3. Secondary Outcome: Occurrence of Seizure With a Start Time >10 Minutes After Administration of the Double-blind Dose
Description: Occurrence of next seizure with a start time >10 minutes and up to 24 hours after administration of the double-blind dose in the CP. Participants who did not have another seizure before the end of the 24-hour observation period were censored at the end of the observation period. Participants administered the open-label second dose who did not have a seizure were censored at the time of the administration.
Time Frame: 24 hours
Population: Randomized participants who received the double-blind dose in the CP.
Measure: Count of Participants; unit: Participants
Arm/Group | USL261 CP | Placebo CP
Number analyzed (Participants) | 134 | 67
Participants | 50 | 31
Statistical Analysis 1: Comparison: USL261 CP vs Placebo CP; Test type: Superiority; p = 0.0124, Log Rank

4. Secondary Outcome: Time to Next Seizure With a Start Time >10 Minutes After Administration of the Double-blind Dose
Description: Time to next seizure with a start time >10 minutes and up to 24 hours after administration of the double-blind dose in the CP. Participants who did not have another seizure before the end of the 24-hour observation period were censored at the end of the observation period. Participants administered the open-label second dose who did not have a seizure were censored at the time of the administration.
Time Frame: 24 hours
Population: Randomized participants who received the double-blind dose in the CP
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | USL261 CP | Placebo CP
Number analyzed (Participants) | 134 | 67
Hours | NA [17.9 to NA] — Median was not estimable as probability of no seizures through 24 hours was above 50%. Upper bound of 95% CI was not estimable. | 12.1 [2.2 to NA] — Upper bound of 95% CI was not estimable.
Statistical Analysis 1: Comparison: USL261 CP vs Placebo CP; Kaplan-Meier estimates; Test type: Superiority; p = 0.0124, Log Rank

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events (TEAEs) collected from administration of first open-label dose of USL261 5 mg in Test Dose Phase (TDP) until completion of the final study visit or 7 days after the last administration of study drug, whichever was later. The duration of individual participant participation was variable as administration of the double-blind dose in the Comparative Phase (CP) was dependent on occurrence of a seizure cluster episode meeting trial criteria after randomization.
Description: Adverse events collected at each visit from participant and/or caregiver. TEAEs presented for TDP and CP separately. Due to the short systemic half-life of active (midazolam), TEAEs within 2 days after administration of first open-label USL261 5 mg dose presented for TDP, and within 2 days after administration of double-blind dose for CP.
Groups:
- USL261 CP, USL261 5 mg Only: Participants completing TDP who received USL261 5 mg as randomized dose to treat a seizure cluster episode in the Comparative Phase (CP)
- USL261 CP, USL261 5 mg + 5 mg: Participants completing TDP who received USL261 5 mg as randomized dose to treat a seizure cluster episode and received an open-label USL261 5 mg dose in the Comparative Phase (CP)
- Placebo CP, Placebo Only: Participants completing TDP who received Placebo as randomized dose to treat a seizure cluster episode in the Comparative Phase (CP)
- Placebo CP, Placebo + USL261 5 mg: Participants completing TDP who received Placebo as randomized dose to treat a seizure cluster episode and received an open-label USL261 5 mg dose in the Comparative Phase (CP)
Arm/Group | USL261 TDP | USL261 CP, USL261 5 mg Only | USL261 CP, USL261 5 mg + 5 mg | Placebo CP, Placebo Only | Placebo CP, Placebo + USL261 5 mg
All-Cause Mortality (participants affected / at risk) | 0/292 | 0/91 | 0/43 | 0/26 | 0/41
Serious Adverse Events (participants affected / at risk) | 2/292 | 0/91 | 0/43 | 0/26 | 1/41
Other Adverse Events (participants affected / at risk) | 78/292 | 17/91 | 10/43 | 3/26 | 7/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | USL261 TDP (N=292) | USL261 CP, USL261 5 mg Only (N=91) | USL261 CP, USL261 5 mg + 5 mg (N=43) | Placebo CP, Placebo Only (N=26) | Placebo CP, Placebo + USL261 5 mg (N=41)
Sedation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure cluster (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | USL261 TDP (N=292) | USL261 CP, USL261 5 mg Only (N=91) | USL261 CP, USL261 5 mg + 5 mg (N=43) | Placebo CP, Placebo Only (N=26) | Placebo CP, Placebo + USL261 5 mg (N=41)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 47 (61) | 5 (5) | 7 (8) | 2 (2) | 3 (3)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 28 (30) | 9 (9) | 4 (4) | 1 (1) | 4 (4)
Lacrimation increased (Eye disorders) | 20 (26) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Product taste abnormal (General disorders) | 17 (19) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 6 (6) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A manuscript or abstract should not be submitted by investigator(s) for publication or presentation until a New Drug Application is approved by the US FDA or permission is granted in writing by sponsor.

DOCUMENTS (2):
  • Study Protocol (2015-05-20): https://cdn.clinicaltrials.gov/large-docs/20/NCT01390220/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-14): https://cdn.clinicaltrials.gov/large-docs/20/NCT01390220/SAP_001.pdf